CLINICAL TRIAL: NCT06929234
Title: Effects of Peer-Supported Health Education on Knowledge, Attitude and Screening for Cervical Cancer in Women: A Mixed Method Randomized Controlled Pilot Study
Brief Title: Effects of Health Education on Knowledge, Attitude and Screening for Cervical Cancer in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Assoc. Prof. Dr., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OrduA2
Record Dates: First submitted 2025-03-21; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Peer Support; Health Education; Cervical Cancers
Keywords: Peer Support; Cervical Cancer; Health; Education
MeSH Terms: conditions — Health Education; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This research will be applied as a "mixed method randomized controlled experimental study". Exploratory sequential mixed design will be used in the study. Quantitative data will be collected first and then qualitative data will be collected.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer-Supported Health Education Group (Experimental): This group will participate in peer-supported health education.
  Interventions: Other: Peer-Supported Health Education
- Basic Health Education Group (Other): This group will participate in basic health education.
  Interventions: Other: Basic Health Education

INTERVENTIONS:
Other: Peer-Supported Health Education — Peer-supported health education will be provided to paticipants in 1 session for an average of 60 minutes in a suitable classroom. In this session, health education will be provided by the researchers and the peer will support the health education. The peer will share her experiences about each part of the training content with the target group in line with the guidance of the researchers, answer questions and make a motivational speech for screening.
  Arms: Peer-Supported Health Education Group
Other: Basic Health Education — What is cervical cancer, what is the importance of cervical cancer, what are the risk factors for cervical cancer, what are the symptoms of cervical cancer, how to screen for cervical cancer, where to get cervical cancer screenings. Participants will be given health education with a power point presentation in a suitable classroom for an average of 45-50 minutes in 1 session.
  Arms: Basic Health Education Group

SUMMARY:
Women's knowledge, attitudes and behaviors about cancer are very important in the prevention of cervical cancer. In addition to medical interventions, psychosocial support and education programs are of great importance in the fight against cancer. Peer support helps individuals going through the same disease process to exchange information and emotional support by sharing their experiences with each other. In addition, the information obtained through peer support provides more permanent learning in individuals due to the transfer of information based on similar experiences and the creation of more trust and empathy compared to traditional education methods. Peer-supported education programs for women diagnosed with cervical cancer not only provide theoretical knowledge but also support the applicability of this knowledge in daily life. The trainings address topics such as risk factors of cervical cancer, the importance of HPV vaccination, the necessity of regular screening tests and healthy lifestyle behaviors, including attitudes towards cervical cancer prevention and cancer-related information. It is very important that this information is not limited to individual learning and that it is discussed within the group and supported by experiences through peer support, in order to increase the level of knowledge.

DETAILED DESCRIPTION:
Detection of cervical cancer at an early stage significantly increases treatment success rates and the quality of life of individuals. Women's knowledge, attitudes and behaviors about cancer are very important in the prevention of cervical cancer. It has been found that the incidence of cervical cancer has decreased in most societies with high levels of awareness about cancer screening. In addition to medical interventions, psychosocial support and education programs are of great importance in the fight against cancer. Peer support helps individuals going through the same disease process to exchange information and emotional support by sharing their experiences with each other. Peer support groups can influence participants' attitudes towards health behaviors by reducing their fear and anxiety about cancer. For women diagnosed with cervical cancer, peer support can facilitate access to accurate information about cancer and help eliminate wrong health behaviors. In this process, women can better understand the importance of participating in screening programs and improve their attitudes towards early diagnosis and preventive health behaviors. In addition, peer-supported information provides more permanent learning in individuals due to the transfer of knowledge based on similar experiences and the creation of more trust and empathy compared to traditional education methods. The effectiveness of education programs increases significantly when they are designed in accordance with the needs and cultural characteristics of the participants. Peer-supported education programs for women diagnosed with cervical cancer not only provide theoretical knowledge but also support the applicability of this knowledge in daily life. The trainings address topics such as risk factors of cervical cancer, the importance of HPV vaccination, the necessity of regular screening tests and healthy lifestyle behaviors, including attitudes towards cervical cancer prevention and cancer-related information. It is very important that this information is not limited to individual learning and that it is discussed within the group and supported by experiences through peer support, in order to increase the level of knowledge. It is important for the effectiveness of the trainings that the individuals providing peer support have sufficient health knowledge about cancer prevention, understand women's health needs and sociocultural norms, speak the same language as women, and are willing to serve as peer supporters. Women who receive peer support share their experiences with screening tests and help other participants learn more about these tests. This increases individuals' trust in health services and encourages them to engage in preventive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled at the Training Center,
* Women between the ages of 30 and 65,
* Women who are married,
* Women who have not been screened for cervical cancer in accordance with the year interval,
* Women who are open to communication and collaboration,
* Women who volunteer to participate in the study will be included in the research.

Exclusion Criteria:

* Women who have had a total hysterectomy,
* Pregnant women,
* Women diagnosed with cervical cancer,
* Women who are screened on time will be excluded from the research.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this study included educations on cervical cancer, the participants will be women.
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Cervical Cancer Knowledge Scale | At baseline and after 4 weeks
  Cervical Cancer Knowledge Scale developed by Haward et al. (2022) was adapted into Turkish by Ergöz Aksoy and Bilgiç (2024). The scale consisted of 8 items and a triple Likert-type rating was used. The items in the scale are evaluated with statements such as True, False, I don't know. In the scoring of the scale, correct answers are worth one point and a maximum of 8 correct answers can be given, so the total score of the scale varies between 0-8. The higher the score obtained from the scale, the higher the knowledge level of the individual. Since the probability of giving a correct answer when guessing a "true or false" item is 50%, participants were allowed to answer "I don't know" to prevent random guesses. In the validity and reliability study of this scale in Turkey, Cronbach's alpha coefficient was found to be 0.80 (Ergöz Aksoy & Bilgiç, 2024).
Attitude Scale for Protection From Cervical Cancer | At baseline and after 4 weeks
  Attitude Scale for Cervical Cancer Prevention developed by Dadak and Koyun in 2017 consists of three sub-dimensions and 22 items. The scale includes ten items for the cognitive sub-dimension, five items for the affective sub-dimension, and seven items for the behavioral sub-dimension. Likert-type rating was used in the scale and the items are evaluated with five statements as (1) Strongly disagree, (2) Somewhat agree, (3) Moderately agree, (4) Mostly agree, (5) Strongly agree. The highest score that can be obtained from the scale is 110 and the lowest score is 22. A high score on the scale indicates that the individual has high attitudes towards prevention of cervical cancer. The Cronbach's Alpha reliability coefficient of the scale was 0.87; the Cognitive sub-dimension was 0.91; the Affective sub-dimension was 0.80 and the Behavioral sub-dimension was 0.84 (Dadak & Taştekin Ouyaba, 2021).

IPD SHARING:
Plan to Share IPD: No